CLINICAL TRIAL: NCT05505513
Title: Can an Array of Micro-electrodes Implanted in a Human Nerve Record Neural Signals and Provide Sensory Feedback Useful for Controlling a Prosthetic Device?
Brief Title: Can an Array of Micro-electrodes Implanted in a Human Nerve Record Neural Signals and Provide Feedback?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, Principle Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 124231
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Amputation
Keywords: Micro-Electrodes; Amputation; Prosthetic Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Implantation of a percutaneous Utah Slanted Electrode Arrays (pUSEAs) (Experimental): The arm (s) of the patient which has been amputated. Intervention include insertion of the percutaneous Utah Slanted Electrode Arrays which will interact with nerve endings in order to gain knowledge about device feasibility and nerve stimulation.
  Interventions: Device: percutaneous Utah Slanted Electrode Arrays (pUSEAs)

INTERVENTIONS:
Device: percutaneous Utah Slanted Electrode Arrays (pUSEAs) — Microelectrode slanted arrays with a large number of electrodes will be surgically implanted into peripheral nerves of patients with limb amputations.

SUMMARY:
The investigators will investigate the device feasibility of human peripheral nerves and muscles recording and stimulation using percutaneous Utah Slanted Electrode Arrays (pUSEAs) implanted into residual peripheral arm nerves and EMG electrodes implanted in the residual muscles of patients with limb amputations in order to determine the ability of the HAPTIX (Hand Proprioception and Touch Interfaces) System to control an upper-extremity prosthesis, and to provide a sense of cutaneous touch and muscle proprioceptive feedback to the amputee.

DETAILED DESCRIPTION:
The investigators will assess the functional capability of microelectrode slanted arrays with a large number of electrodes implanted into peripheral nerves of patients with upper-limb transradial amputations. The investigators hypothesize that recording neural signals from individual electrodes will provide selective motor information that is adequate to allow control over artificial limbs with many moving parts, i.e., wrist, and individually moving digits. These studies will also investigate to what extent microstimulation can provide sensory feedback from a prosthetic limb.

The HAPTIX System study will investigate the safety and efficacy of using electromyography (EMG), plus neural recording and nerve stimulation, to control and provide cutaneous and proprioceptive feedback from a dexterous, motorized and sensorized, upper-extremity prosthesis (e.g., the DEKA LUKE arm) used by amputees.

The HAPTIX System is intended to permit the function of an upper-extremity prosthesis to assist in activities of daily living (ADLs) using neurostimulation and recording of EMG and neural signals to control the prosthesis, and evoke touch sensation and proprioception in upper-extremity amputees with DEKA LUKE sensorized upper extremity prosthesis.

The HAPTIX System study is an early feasibility study (EFS) of the use of a combination of EMG recording electrodes, neural recording and stimulating electrodes, and external electronics and algorithms designed to provide sensory and proprioceptive feedback to the amputee, and to control movements of a prosthetic hand.

EMG signals from the residual forearm muscles of amputees will be recorded using up to 8 custom bipolar PermaLoc® electrodes. The incorporation of these electrodes into the HAPTIX System is described in 001_G190131A002_Amended_Device Description. Nerve signals will also be recorded using up to 3 percutaneous Utah Slanted Electrode Arrays (pUSEAs), whose electrode tips will be implanted intrafascicularly in residual arm nerves. Present-version pUSEAs utilize a transcutaneous lead and extracorporeal connector. Motor signals from the nerve will contribute to decoding motor intents decoded to control an advanced prosthetic hand. Nerve stimulation to evoke sensory perceptions will be provided by passing current through individual pUSEA electrodes, separately or in combination.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age and less than 65 years of age
* unilateral and bilateral traumatic or elective upper extremity amputations at the transradial level

Exclusion Criteria:

* incarceration
* pregnancy
* inability to consent
* psychiatric comorbidity
* medical conditions that significantly increase the risk of adverse effects of general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measure Action Potentials (millivolts, mV) | Up to 2-years Follow-up
  Three participants after receiving a stimuli will have action potentials (millivolts, mV) arising from the axons surrounding the tip of each electrode recorded in time. The moving action potentials (mV) measure five phases: resting potential, depolarization, peak, repolarization, and hyperpolarization.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hutchinson, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- The University Orthopaedic Center, Salt Lake City, Utah, United States